CLINICAL TRIAL: NCT02777333
Title: Simulation-based Arthroscopic Surgery Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MSD-IDREC-C1-2014-152
Record Dates: First submitted 2016-05-10; First posted 2016-05-19 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2016-05

CONDITIONS: Arthroscopy Training
Keywords: Simulation; Arthroscopy; Motion analysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simulation training (Experimental): Addition of simulation training during usual clinical training as part of a GMC (General Medical Council) recognised Deanery training programme
  Interventions: Behavioral: Simulation training
- Non-simulation/Routine training (No Intervention): Usual clinical training as part of a GMC (General Medical Council) recognised Deanery training programme

INTERVENTIONS:
Behavioral: Simulation training — Simulation training in a skills lab for 1 hour per week over 13 weeks on dry, bench-top box trainers and anatomical simulators
  Arms: Simulation training

SUMMARY:
The purpose of this study is to determine whether simulation training improves the performance during arthroscopic surgery ('keyhole' surgery into a joint).

DETAILED DESCRIPTION:
This single blinded randomised controlled study of junior orthopaedic trainees aims to assess whether the addition of simulation training improves arthroscopic technical skills performance of junior orthopaedic trainees during knee arthroscopy in the operating theatre compared to their usual clinical training programme. This will be assessed using objective motion analysis parameters recorded from wireless elbow-mounted motion sensors during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Healthy adults, Male or Female, aged 18 years or above.
* Enrolled in Health Education Thames Valley/Oxford Deanery Training Programme in junior surgical training posts

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Previously completed higher surgical training programme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L Rees, FRCS-Tr&Orth, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SHO trainees (PGY 2-3 equivalent) within nationally approved T&O training rotations at an English teaching hospital were eligible for inclusion. Exclusions; more than 2 years of surgical training; previous admission to a higher surgical training program; performed or assisted in over 10 arthroscopic or minimal-access procedures.
Period: Overall Study
Arm/Group | Simulation Training | Non-simulation/Routine Training
Started | 15 | 15
Completed | 15 | 13
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Simulation Training: Addition of simulation training during usual clinical training as part of a GMC (General Medical Council) recognised Deanery training programme Simulation training: Simulation training in a skills lab for 1 hour per week over 13 weeks on dry, bench-top box trainers and anatomical simulators
- Total: Total of all reporting groups
Arm/Group | Simulation Training | Non-simulation/Routine Training | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 26.02 [25.76 to 27.18] | 26.34 [26.09 to 27.17] | 26.18 [25.76 to 27.18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 7 | 9 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Postgraduate year [Count of Participants; unit: Participants]
  PGY2 | 12 | 12 | 24
  PGY3 | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Hand Movements Required by Participants to Perform a Diagnostic Arthroscopy of the Knee in Theatre
Description: Wireless elbow-mounted accelerometer and gyroscopic sensors worn by the participant will generate 6 degree of freedom motion data (three rotational degrees around the x, y and z axes, known as 'roll', 'pitch', and 'yaw', and three translational degrees of freedom along x, y and z axes, known as 'surge', 'sway' and 'heave') which will be analysed using validated, bespoke algorithms to calculate the number of hand movements taken whilst performing a diagnostic knee arthroscopy according to a standardised protocol.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: hand movements
Arm/Group | Simulation Training | Non-simulation/Routine Training
Number analyzed (Participants) | 15 | 13
hand movements | 544 [465 to 593] | 893 [747 to 1242]

2. Secondary Outcome: Smoothness of Hand Movements by Participants to Perform a Diagnostic Arthroscopy of the Knee in Theatre
Description: Wireless elbow-mounted accelerometer and gyroscopic sensors worn by the participant will generate 6 degree of freedom motion data which will be analysed using validated, bespoke algorithms to calculate the smoothness (also known as 'jerk', the first derivative of acceleration by time, or third derivative of distance by time) of hand movements taken whilst performing a diagnostic knee arthroscopy according to a standardised protocol according to a standardised protocol.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: ms^-3
Arm/Group | Simulation Training | Non-simulation/Routine Training
Number analyzed (Participants) | 15 | 13
ms^-3 | 25,842 [20,867 to 27,468] | 36,846 [29,840 to 53,949]

3. Secondary Outcome: Time Taken by Participants to Perform a Diagnostic Arthroscopy of the Knee in Theatre
Description: Wireless elbow-mounted accelerometer and gyroscopic sensors worn by the participant will generate 6 degree of freedom motion data which will be analysed using validated, bespoke algorithms. These data will also collect time signatures, which can be used to work out the time taken by participants to perform a diagnostic arthroscopy of the knee in theatre according to a standardised protocol.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Simulation Training | Non-simulation/Routine Training
Number analyzed (Participants) | 15 | 13
seconds | 320 [294 to 392] | 573 [477 to 860]

4. Secondary Outcome: Minor Hand Movements Required by Participants to Perform a Diagnostic Arthroscopy of the Knee in Theatre
Description: Wireless elbow-mounted accelerometer and gyroscopic sensors worn by the participant will generate 6 degree of freedom motion data (three rotational degrees around the x, y and z axes, known as 'roll', 'pitch', and 'yaw', and three translational degrees of freedom along x, y and z axes, known as 'surge', 'sway' and 'heave') which will be analysed using validated, bespoke algorithms to calculate the number of movements (below the threshold for 'hand movements' above in outcome 1, but above the data noise threshold) taken whilst performing a diagnostic knee arthroscopy according to a standardised protocol.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: minor hand movements
Arm/Group | Simulation Training | Non-simulation/Routine Training
Number analyzed (Participants) | 15 | 13
minor hand movements | 176 [133 to 209] | 435 [310 to 652]

5. Secondary Outcome: Stationary Time of Participants to Perform a Diagnostic Arthroscopy of the Knee in Theatre
Description: Wireless elbow-mounted accelerometer and gyroscopic sensors worn by the participant will generate 6 degree of freedom motion data which will be analysed using validated, bespoke algorithms. These data will also collect time signatures, which can be used to work out the length of time during the procedure where each hand is stationary while participants perform a diagnostic arthroscopy of the knee in theatre according to a standardised protocol.
Time Frame: 3 months
Population: Data were not collected
Arm/Group | Simulation Training | Non-simulation/Routine Training
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Idle Time of Participants to Perform a Diagnostic Arthroscopy of the Knee in Theatre
Description: Wireless elbow-mounted accelerometer and gyroscopic sensors worn by the participant will generate 6 degree of freedom motion data which will be analysed using validated, bespoke algorithms. These data will also collect time signatures, which can be used to work out the length of time during the procedure where both hands are stationary at the same time while participants perform a diagnostic arthroscopy of the knee in theatre according to a standardised protocol.
Time Frame: 3 months
Population: Data were not collected
Arm/Group | Simulation Training | Non-simulation/Routine Training
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Dominance of Participants to Perform a Diagnostic Arthroscopy of the Knee in Theatre
Description: Wireless elbow-mounted accelerometer and gyroscopic sensors worn by the participant will generate 6 degree of freedom motion data which will be analysed using validated, bespoke algorithms. These data will be analysed for the relative activity and dominance of each hand during the procedure while participants perform a diagnostic arthroscopy of the knee in theatre according to a standardised protocol.
Time Frame: 3 months
Reporting Status: Not Posted

8. Secondary Outcome: Global Rating Scale Performance During Diagnostic Knee Arthroscopy in Theatre
Description: Validated global rating scale for assessing diagnostic knee arthroscopy performance
Time Frame: 3 months
Population: Data were not collected
Arm/Group | Simulation Training | Non-simulation/Routine Training
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Deviation From 'Idealised' Motion Parameters for Participants to Perform a Diagnostic Arthroscopy of the Knee in Theatre
Description: Previously described motion parameters of participants performing a diagnostic knee arthroscopy in theatre (see Primary outcome 1, and secondary outcomes 2-8) reported as a ratio to the 'ideal' performance as measured from the supervising clinician performing an optimal diagnostic knee arthroscopy on the same patient as the participant while wearing the wireless elbow-mounted accelerometer and gyroscopic sensors which will record 6 degree of freedom motion data to allow calculation of 'number of hand movements', 'smoothness', 'time taken', 'minor hand movements', 'stationary time', 'idle time' and dominance'
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: Performance ratio (Participant:superviso
Arm/Group | Simulation Training | Non-simulation/Routine Training
Number analyzed (Participants) | 15 | 13
Performance ratio (Participant:superviso
  Ratio of Hand movements | 1.9 [1.5 to 2.1] | 3.3 [2.2 to 4.8]
  Ratio of Minor hand movements | 3.8 [2.8 to 4.7] | 10.3 [5.1 to 11.9]
  Ratio of Smoothness | 1.2 [1.1 to 1.7] | 2.6 [1.6 to 3.0]
  Ratio of Time taken | 2.1 [1.8 to 2.8] | 4.3 [2.8 to 5.4]

10. Secondary Outcome: Motion Analysis Parameters During Simulation
Description: Change in participant performance on dry, bench top box trainers and anatomical simulators between baseline and 3 months using motion analysis parameters described in Primary outcome 1 and secondary outcomes 2-8 as measured by wireless elbow-mounted accelerometer and gyroscopic sensors
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: Hand movements
Arm/Group | Simulation Training | Non-simulation/Routine Training
Number analyzed (Participants) | 15 | 15
Hand movements | 131 [108 to 153] | 249 [197 to 345]

11. Secondary Outcome: Resting State Network Functional Changes on fMRI (Functional Magnetic Resonance Imaging)
Description: Use of MELODIC (Multivariate Exploratory Linear Optimized Decomposition into Independent Components) to identify resting state networks, and analyse differences in functional connectivity at baseline and three months between the intervention and control arms.
Time Frame: 3 months
Reporting Status: Not Posted

12. Secondary Outcome: Voxel Based Morphometry Structural Changes on fMRI (Functional Magnetic Resonance Imaging)
Description: Using FSLVBM (fMRIB's Software Library Voxel Based Morphometry) to calculate voxel-wise changes in grey matter volumes at baseline and three months between the intervention and control arms. Changes in VBM imply changes in grey matter volume and represent structural brain change.
Time Frame: 3 months
Reporting Status: Not Posted

13. Secondary Outcome: Diffusion Tractography Structural Changes on fMRI (Functional Magnetic Resonance Imaging)
Description: Using FDT (fMRIB's Diffusion Toolbox) to model local diffusion and changes in tractography at baseline and three months between the intervention and control arms. Changes in diffusion imply micro-structural (axonal) connectivity and represent structural brain change.
Time Frame: 3 months
Reporting Status: Not Posted

14. Secondary Outcome: Quantitative Magnetisation Transfer Structural Changes on fMRI (Functional Magnetic Resonance Imaging)
Description: Quantitative magnetisation transfer imaging estimates liquid and semisolid (macromolecular) constituents of tissue at baseline and three months between the intervention and control arms. Changes in macromolecular content imply micro-structural (myelin) connectivity and represent structural brain change.
Time Frame: 3 months
Reporting Status: Not Posted

15. Secondary Outcome: Feasibility of Additional Simulation Training
Description: Qualitative survey of participants opinions of the addition of simulation to their usual clinical training programme
Time Frame: 3 months
Population: Data were not collected
Arm/Group | Simulation Training | Non-simulation/Routine Training
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks (study period)
Arm/Group | Simulation Training | Non-simulation/Routine Training
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Some outcomes were not analysed as stated in the trial protocol as during the construct validation stage these were found to not correlate with performance

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT02777333/Prot_SAP_000.pdf